CLINICAL TRIAL: NCT03612323
Title: Comparative Evaluation of the Efficacy of Intra-ligamentary Injection of 20 Milligram (Mg) Piroxicam Versus 4% Articaine in Management of Endodontic Pain in Patients With Symptomatic Irreversible Pulpitis in Mandibular Molars
Brief Title: Comparison Between Intraligamentary Piroxicam and Articaine
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lobna Elhadad, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Piroxicam_Articaine
Record Dates: First submitted 2018-07-16; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — Piroxicam; Carticaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-ligamentary Piroxicam (Experimental): Piroxicam is a long acting potent Non steroidal anti-inflammatory drug (NSAID)with half life of 50 hours in plasma, is given as intervention to assess the pain,will be administered by intra-ligamentary technique by injecting 0.4 milliliter (mL) of 20 milligram (Mg) piroxicam.
  Interventions: Drug: Intra-ligamentary Piroxicam
- Intra-ligamentary Articaine (Active Comparator): Articaine is a local anesthetic agent, will be administered by intraligamentary technique by injecting 0.4 milliliter (mL) of 4% articaine
  Interventions: Drug: Intra-ligamentary Articaine

INTERVENTIONS:
Drug: Intra-ligamentary Piroxicam — Piroxicam is a long-acting potent analgesic non selective oxicams derivative, has a half-life of 50 hrs in the plasma.The onset of action of oral piroxicam is 2-4 hrs, but it is anticipated that injectable piroxicam could produce more rapid onset of action. It could favourably overcome the intense pain up to 48 hrs following the treatment
  Other Names: Feldene
  Arms: Intra-ligamentary Piroxicam
Drug: Intra-ligamentary Articaine — Articaine is a local anesthetic agent , has been reported to be an effective anesthetic in controlling pain during root canal treatment
  Other Names: Articaine
  Arms: Intra-ligamentary Articaine

SUMMARY:
Comparing the efficacy of intra-ligamentary Piroxicam and intra-ligamentary Articaine on pain during and after endodontic treatment of mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Owing to the painful nature of endodontic treatment in teeth with symptomatic irreversible pulpitis and difficulty in achieving effective anesthesia particularly in mandibular molars due to various factors such as different bony landmarks, anatomical variations, needle deflection, accessory innervation, so local anesthesia isn't enough in such cases. Piroxicam is a long-acting potent analgesic non selective oxicams derivative, has a half-life of 50 hrs in the plasma.The onset of action of oral Piroxicam is 2-4 hrs, but it is anticipated that injectable piroxicam could produce more rapid onset of action. It could favourably overcome the intense pain up to 48 hrs following the treatment. It is also postulated that the intraligamentary injection enables the application of anti-inflammatory agents in the periapical intraosseous region. Moreover, intra-ligamentary injection of local anesthesia was reported to be an effective and easy way to control severe pain during endodontic treatment mainly in mandibular teeth which are more difficult than maxillary teeth , thus piroxicam may be effective as an adjuvant drug to support the action of local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and medically free patients.
* Acute symptomatic irreversible pulpitis of the mandibular first or second molar teeth.
* Vital teeth with no history of previous root canal treatment.
* Teeth that could be treated endodontically in single visit.
* Teeth with normal periodontium, not sensitive to percussion with no periapical radiolucency.
* Patients able to understand numerical rating scale and sign the informed consent.

Exclusion Criteria:

* Known hypersensitivity to piroxicam.
* Pregnancy or lactation.
* Asthma or allergy to other anti-inflammatory drugs.
* History of peptic ulceration.
* Teeth associated with swelling or fistulous tract, acute or chronic periapical abscess.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Alleviation of post-operative pain severity | up to 48 hours
  the patient will be asked to rate the progress of pain on the NRS and inform the investigator with the results,Primary outcome will be collected by the operator through Numerical Rating Scale (NRS) which is an 11-point scale consisting of numbers from 0 through 10; 0 reading represents "no pain" , 1- 3 readings represent "mild pain" , 4- 6 readings represent "moderate pain" , 7- 10 readings represent "severe pain" No or mild pain will be considered as success while moderate or severe pain will be regarded as failure.

SECONDARY OUTCOMES:
Intra-operative pain during access cavity preparation and instrumentation which will be measured ny Numerical Rating Scale (NRS) | immediately after injection of the drug up to 2 hours till end of endodontic treatment
  the patient will be asked to rate the progress of pain on the NRS and inform the investigator with the results,secondary outcome will be assessed through Numerical Rating Scale (NRS) which is an 11-point scale consisting of numbers from 0 through 10; 0 reading represents "no pain" , 1- 3 readings represent "mild pain" , 4- 6 readings represent "moderate pain" , 7- 10 readings represent "severe pain" No or mild pain will be considered as success while moderate or severe pain will be regarded as failure.

CONTACTS AND LOCATIONS:
Overall Officials: Lobna Elhadad, Student, Principal Investigator — Cairo University